CLINICAL TRIAL: NCT07061184
Title: The Efficacy of Fengliao Changweikang Keli for Patients With Diarrhea-predominant Irritable Bowel Syndrome: Study Protocol for a Multicenter, Randomized, Placebo-controlled N-of-1 Trial
Brief Title: Fengliao Changweikang for Diarrhea-predominant Irritable Bowel Syndrome: N-of-1 Trial
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, DONG WU, Chief physician of Gastroenterology, Peking Union Medical College Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: I-25PJ1478; 2022YFC2504006 (Other Grant/Funding Number: Ministry of Science and Technology, China)
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Irritable Bowel Syndrome - Diarrhoea; Traditional Chinese Medicine (TCM); N of 1 Study Design; Efficacy and Safety

STUDY DESIGN:
Intervention Model Description: N-of-1 trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FLCWK (Experimental): FLCWK one sachet (8 g) to be taken three times daily in 1 month treatment peroid, 3 treatment periods in 9 months
  Interventions: Drug: FLCWK; Drug: Placebo
- Placebo (Placebo Comparator): Placebo one sachet (8 g) to be taken three times daily in 1 month treatment peroid, 3 treatment periods in 9 months
  Interventions: Drug: FLCWK; Drug: Placebo

INTERVENTIONS:
Drug: FLCWK — FLCWK and matching placebo to be taken in a randomised order for 9 months
Drug: Placebo — FLCWK and matching placebo to be taken in a randomised order for 9 months

SUMMARY:
Irritable bowel syndrome with diarrhea (IBS-D) is a functional gastrointestinal disorder, with characteristics of defecation related abdominal pain and diarrhea. Routine treatment strategy for IBS-D is symptom-based with unsatisfactory results, while there is a growing interest in complementary and alternative medicine such as Traditional Chinese Medicine. However, lack of high-quality evidences being the obstacle for its development.

This study aims to evaluate the efficacy of Fengliao Changweikang Keli (FLCWK) on symptoms and health-related quality of life in mild to moderate IBS-D patients.

After 2-week run-in period, each participant will be randomized to a sequence of six 4-week double-blind treatment periods of FLCWK 8 g three times daily or placebo, separated by 2-week washout periods.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 75 years.
2. Mild to moderate IBS-D patients, with IBS Severity Scoring System (IBS-SSS) scores of 75 to 300 points[14].
3. Ability to complete questionnaires and provide written informed consent.
4. Current use of IBS medications (probiotics, antibiotics, antispasmodic, antidiarrheal and neuromodulators) should be prescribed on a stable dose at least 30 days prior to enrollment, and have no plan to change the dose, diet or lifestyle.
5. Normal blood cell count, liver function, creatinine and urea levels within the last 2 weeks.

Exclusion Criteria:

1. History of organic gastrointestinal diseases such as inflammatory bowel disease, celiac disease and malignancy.
2. Scores of IBS-SSS > 300 points or IBS-SSS < 75 points.
3. History of severe heart, kidney or liver diseases.
4. Pregnant or breastfeeding.
5. Current alcohol or drug abuse.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
IBS-SSS score | At the end of run-in period (week 2) and at the end of each washout period (week 8, 14, 20, 26, 32) and during each treatment period (week 6, 12, 18, 24, 30, 36).
  The severity score questionnaire consists of 5 items and each item is rated on a scale of 0-100 points, leading to a total score of 0-500 points. An improvement of more than 50 points for IBS-SSS questionnaire is considered clinical effective.

SECONDARY OUTCOMES:
IBS-QOL score | At the end of run-in period (week 2) and at the end of each washout period (week 8, 14, 20, 26, 32) and during each treatment period (week 6, 12, 18, 24, 30, 36).
  IBS-QOL is a 34-item questionnaire assessing patient's health related quality of life, and higher scores indicate a better quality of life. IBS-QOL focuses on eight domains, namely dysphoria, activity interference, body image, health worry, food avoidance, social reaction, sexual and relationships, and an increase of more than 14 points indicates clinical improvement in quality of life. The minimal clinically important difference (MCID) on the IBS-QOL is defined as a change of 10 points in the total score.
self-reported symptoms including abdominal pain and diarrhea | At the end of run-in period (week 2) and at the end of each washout period (week 8, 14, 20, 26, 32) and during each treatment period (week 6, 12, 18, 24, 30, 36).
  The score of worst abdominal pain in the past 24 hours will be evaluated by visual analogue scale (VAS) ranging from 0 to 10. The stool consistency of the past 24 hours will also be rated by BSFS, based on a 1 to 7 scale where 1 corresponds to a hard stool and 7 corresponds to watery diarrhea.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No